CLINICAL TRIAL: NCT01316705
Title: COMPARISON BETWEEN IMSI AND ICSI TECHNIQUES WITH DONATED EGGS
Brief Title: Comparison Between Intracytoplasmic Morphologically Selected Sperm Injection (IMSI) And Intra Cytoplasmic Sperm Injection (ICSI) Techniques With Eggs Donated
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Manuela Alonso, Biologist, IVI Madrid
Other Study IDs: MAD-MA-11-2009-02
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Sperm Head

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to determine if early embryonic development, in D2 and D3 and the blastocyst, is compromised by the fine morphology of sperm nucleus. This will draw the IMSI, in which sperm will be chosen using the classification MSOME and ICSI in which sperm morphology is elected with less magnification. Both techniques are performed in oocytes of donor , being the coohorte used for both techniques picked at random. All courses will begin as a crop sequence, using the criteria of the IVF laboratory. Transfers will be made in blastocyst stage (D5 or D6), except in cases where the number of fertilized is less than 6 or fewer than 6 embryos of acceptable quality in D3, which would transfer the same D3 . With donor oocytes, the quality of these need not be compromised and to perform the same technique in all oocytes results in pure transfers with both techniques. It allows us to compare results in term of pregnancy, implantation and early abortion rate, as well as embryo quality.

DETAILED DESCRIPTION:
ICSI is the most frequent insemination method used at all IVI clinics. This technique allows the observation of both, oocytes and spermatozoa, at a maximum magnification of 400X. At this magnification we are only able to assess gross morphological characteristics such as: double heads, double tails, globozoospermia, megalozoospermia.

Nowadays, many groups are using a new method to select spermatozoa known as MSOME (high magnification motile sperm organelle morphology examination) (Bartoov B, et al.,2002). This method allows us to perform a fine assessment of the sperm nucleus and to select at a very high magnification and in real time. The magnification used is between 600 and 13500x.

Later the group of Bartoov introduced the IMSI (intracytoplasmic morphologically selected sperm injection) (Bartoov B., et al., 2003), allowing the single microinjection of selected motile spermatozoa with strictly defined morphologically normal nuclei into the cytoplasm of retrieved oocytes. This prospective controlled study, performed in couples with male infertility and at least two previous failed ICSI attempts, showed that IMSI resulted in a significantly higher pregnancy and implantation rate as compared with conventional ICSI. From their results they assume that in the IMSI, the survival of the embryo in the uterus is associated with the fine morphological state of the sperm nucleus.

Following these data have been some groups, such as Antinori M. et al., 2007, or Vanderzwalmen P et al., 2007 and 2008, showing spectacular results in pregnancy and implantation rate with this new technique, in couples who had several unsuccessful cycles of assisted reproduction. One objection of this work is that all comparisons have been made by relating the results of the IMSI with retrospective results of previous cycles of ICSI.

This study aims to determine if early embryonic development, in D2 and D3 and the blastocyst, is compromised by the fine morphology of sperm nucleus. This will draw the IMSI, in which sperm will be chosen using the classification MSOME and ICSI in which sperm morphology is elected with less magnification. Both techniques are performed in oocytes of donor , being the coohorte used for both techniques picked at random. All courses will begin as a crop sequence, using the criteria of the IVF laboratory. Transfers will be made in blastocyst stage (D5 or D6), except in cases where the number of fertilized is less than 6 or fewer than 6 embryos of acceptable quality in D3, which would transfer the same D3 . With donor oocytes, the quality of these need not be compromised and to perform the same technique in all oocytes results in pure transfers with both techniques. It allows us to compare results in term of pregnancy, implantation and early abortion rate, as well as embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* teratozzospermia in the sperm sample
* more than 9 oocytes (MII)

Exclusion Criteria:

* no egg donation cycles
* less than 10 MII
* vitrified oocytes
* no teratozoospermia males

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: - Egg donation cycles
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)